CLINICAL TRIAL: NCT00677482
Title: Cytomegalovirus (CMV) microRNA Expression in Vivo and Immune Evasion Correlates
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: 7304
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2015-05

CONDITIONS: Transplant
Keywords: liver transplant; lung transplant; kidney transplant; heart transplant; CMV microRNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Solid organ transplant recipients with both asymptomatic CMV viremia, and symptomatic CMV disease are eligible for inclusion in the study. THis includes liver, kidney, heart, pancreas, lung, intestinal and combined transplant recipients.

SUMMARY:
Cytomegalovirus (CMV) is the most common viral infection in patients who have undergone a transplant.Serious infections due to CMV can affect many parts of the body including the lungs, the gut, and the liver. The purpose of this study is to assess how the virus interacts with the patient's immune system, so that in the future it may be possible to develop better ways to prevent and treat the virus infection.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) disease is an important cause of morbidity in solid organ transplantation recipients. Viral reactivation, either of donor origin or endogenous latent virus involves a complex series of steps. A number of factors contribute to the CMV reactivation from latency including exogenous immunosuppression, pre-existing host immunity, and cytokine dysregulation [1,2]. Symptomatic patients are classified as having CMV disease, which presents as a viral syndrome (fever, malaise) or as tissue invasive disease, such as hepatitis or pneumonitis. CMV can also have indirect manifestations due to an immunomodulatory effect of viral replication, resulting in other opportunistic infections and acute and chronic allograft injury [2-4]. CMV disease in organ transplant recipients is generally treated with a finite course of intravenous or oral antiviral therapy. However, the risk of recurrent CMV disease is estimated to be between 25-30% [5-7].

The pathogenesis of CMV reactivation, viral replication, disease progression, and viral persistence is likely related to a number of host factors in transplant patients, including degree and type of immunosuppressive therapy, and pre-existing immunity [8,9]. However, CMV is a remarkably complex virus with a large genome encoding approximately 200 open reading frames. A number of viral factors likely also play a role in determining the risk of CMV disease, the risk of tissue invasion, the response to therapy, and the risk of recurrence once therapy is initiated. The virus commits a large percentage of its total genome coding capacity to the tasks of modulating host cell behaviour and host response to infection [8,9]. These include CMV gene products aimed at escaping host defence mechanisms which are commonly referred to as CMV immune evasion genes [9-11]. Some of these immune evasion genes encode for proteins that can actively interfere with distinct steps in the antigen expression pathway and thus contribute to viral persistence despite an active host immune response. For example US2, US3, US6, and US11 encode for a protein whose ultimate effect is to reduce the levels of MHC class I proteins on the surface of infected cells. The CMV UL141 gene product provides protection against killing by a wide array of NK cell populations, via blocking of surface expression of NK cell-activating ligand CD155 [26]. Also, human CMV expresses several homologues of host G protein-coupled receptors (GPCRs), of which the chemokine receptor homologue US28 is the best characterized [27]. Although the exact significance of US28 has not been determined, the protein product may play a role in cell entry, leukocyte chemotaxis, viral dissemination and immune evasion [27].

MicroRNAs MicroRNAs are recently discovered small endogenous non-coding RNAs. These small RNAs of ~22 nucleotide length are crucial post-transcriptional regulators of gene expression in a wide spectrum of normal and abnormal biological processes including antiviral defence, oncogenesis and development in higher eukaryotes. Recently several virus genomes have also been found to encode microRNAs. The present understanding of the biological functions of virus-encoded microRNAs remains sketchy, with evidence mainly derived from studies on individual or a small set of microRNAs encoded by the viruses and their cognate hosts. Survival strategies of the virus and counter strategies of host cells through miRNAs of host and viral origin and their respective targets form the crux of host virus interactions mediated by microRNAs. Thus microRNAs form a complex link between the regulatory networks of the host and the pathogen. A thorough understanding of the microRNA-mediated host-pathogen interaction is essential in understanding the basic pathophysiological changes associated with viral infections

MicroRNAs and CMV A number of viral microRNAs have been found in CMV. The function of the majority of these is largely unknown. Recently, the function of a specific microRNA (miR-UL-112-1) encoded by CMV was partially elucidated. Stern-Ginossar et al. used a new bioinformatics tool to identify the major histocompatibility complex (MHC) class I-related chain B (MICB) mRNA as a target of a miRNA encoded by CMV. MICB is a cellular ligand for the activating receptor NKG2D, which is expressed on some natural killer cells, γ/δ T cells, and CD8+ T cells. During cellular stress, such as that caused by viral infection, MICB is induced, thus activating natural killer and T cells that can lead to the killing of infected cells. Therefore blocking this process would probably benefit the virus. Stern-Ginossar et al. showed that cells infected with CMV that have been engineered to lack the miR-UL112-1 were more susceptible to being killed in an NKG2D-dependent manner by natural killer cells. The CMV-encoded protein UL16, also provides protection against the detection of infected cells by natural killer cells, by sequestering MICB in the intracellular milieu and preventing it from reaching the cell surface. Why the virus has two different mechanisms to achieve the same goal is not clear, particularly since the closely related NKG2D-ligand MICA is induced during viral infection. Members of my laboratory and I have recently described2 another function of the same miRNA. Successful, persistent infection depends on the maintenance of cell viability despite the production of toxic viral proteins. One way in which CMV can restrict the production of viral proteins is by restricting viral replication. We observed that miR-UL112-1 down-regulates the expression of CMV genes involved in its own replication process, in part by targeting a viral mRNA (encoding a protein called immediate early 72) that regulates the transcription of viral genes required for acute replication.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients who fulfill the following criteria are eligible for inclusion:

* Age >=18 years
* Solid Organ Transplant Recipients
* Documented CMV disease or asymptomatic CMV viremia

Exclusion Criteria:

* Unable to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ tranplant recipients with both asymptomatic CMV viremia and symptomatic CMV disease are eligible for inclusion in the study. This include liver, kidney, heart, pancreas, lung, intestinal and combined transplant recipients.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07-27 (Actual); Study Completion 2013-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Gandhi MK, Khanna R. Human cytomegalovirus: clinical aspects, immune regulation, and emerging treatments. Lancet Infect Dis. 2004 Dec;4(12):725-38. doi: 10.1016/S1473-3099(04)01202-2. PMID 15567122
- [Background] Preiksaitis JK, Brennan DC, Fishman J, Allen U. Canadian society of transplantation consensus workshop on cytomegalovirus management in solid organ transplantation final report. Am J Transplant. 2005 Feb;5(2):218-27. doi: 10.1111/j.1600-6143.2004.00692.x. PMID 15643981
- [Background] Humar A, Kumar D, Boivin G, Caliendo AM. Cytomegalovirus (CMV) virus load kinetics to predict recurrent disease in solid-organ transplant patients with CMV disease. J Infect Dis. 2002 Sep 15;186(6):829-33. doi: 10.1086/342601. Epub 2002 Aug 28. PMID 12198618
- [Background] Rasmussen L. Molecular pathogenesis of human cytomegalovirus infection. Transpl Infect Dis. 1999 Jun;1(2):127-34. doi: 10.1034/j.1399-3062.1999.010206.x. PMID 11428980
- [Background] Tomasec P, Wang EC, Davison AJ, Vojtesek B, Armstrong M, Griffin C, McSharry BP, Morris RJ, Llewellyn-Lacey S, Rickards C, Nomoto A, Sinzger C, Wilkinson GW. Downregulation of natural killer cell-activating ligand CD155 by human cytomegalovirus UL141. Nat Immunol. 2005 Feb;6(2):181-8. doi: 10.1038/ni1156. Epub 2005 Jan 9. PMID 15640804